CLINICAL TRIAL: NCT03496584
Title: Effects of Phytonutrients on Vascular and Skin Health and Systemic Inflammation in Obese Men
Brief Title: Effects of Phytonutrients on Vascular Health and Skin in Obese Males
Acronym: PomSkin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding to complete study
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-001781
Record Dates: First submitted 2018-03-29; First posted 2018-04-12 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Erythema; Inflammation
MeSH Terms: conditions — Erythema; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pomegranate Juice (Active Comparator): Postprandial high fat meal will be administered with pomegranate juice with the first dose of the intervention, Pomegranate Juice , followed by 12 weeks of pomegranate juice consumption.
  Interventions: Other: Pomegranate Juice
- Placebo Juice (Placebo Comparator): Postprandial high fat meal will be administered with pomegranate juice with the first dose of the intervention, Placebo Juice , followed by 12 weeks of pomegranate juice consumption.
  Interventions: Other: Placebo Juice

INTERVENTIONS:
Other: Pomegranate Juice — After the one week run-in period of consuming an ellagitannin-free diet, participants will undergo the skin testing followed by the postprandial meal test with a high fat (HF) test meal consumed with the first dose of the intervention (Pom J or placebo). For the next 12 weeks, participants will consume a daily dose of pomegranate juice 1x/day. During week 4 participants will undergo another skin testing. During week 12 participants will undergo another skin testing and postprandial meal challenge. Stool will be collected at week 1, 4 and 12.
  Arms: Pomegranate Juice
Other: Placebo Juice — After the one week run-in period of consuming an ellagitannin-free diet, participants will undergo the skin testing followed by the postprandial meal test with a high fat (HF) test meal consumed with the first dose of the intervention (Pom J or placebo). For the next 12 weeks, participants will consume a daily dose of placebo juice 1x/day. During week 4 participants will undergo another skin testing. During week 12 participants will undergo another skin testing and postprandial meal challenge. Stool will be collected at week 1, 4 and 12.
  Arms: Placebo Juice

SUMMARY:
This study will determine the effects of beneficial compounds of plant foods, such as pomegranate on cardiovascular health, skin inflammation and aging. This will be tested by asking healthy males to eat a high fat ground beef patty with 8oz. pomegranate juice or 8oz placebo (a study product that looks like pomegranate juice, but contains no active ingredients) and then measuring blood vessel dilation (endothelial function) by blood flow. The investigators also will measure the amount of Nitric Oxide (NO) in blood and urine samples and sugar and insulin in blood. In addition, a Cutometer, a device that measures the elasticity of the skin, will be used to obtain measurements of skin inflammation and aging.

Healthy men have been chosen for this study because eating high fat hamburger patties can easily mimic in them the condition that causes atherosclerosis. The results from this study may help to explain how high fat foods can be harmful to the body and how beneficial plant foods can have on cardiovascular function and the skin.

DETAILED DESCRIPTION:
The proposed investigation has two major objectives: 1. to determine the clinical efficacy of pomegranate juice to reduce skin aging by assessing UV-induced change and skin biological characteristics of elasticity, sebum, hydration/moisture and systemic inflammation and 2. To determine the impact of pomegranate polyphenols on the metabolic response to a high fat meal by postprandial flow-mediated dilation and plasma nitric oxide. The investigators propose to achieve the following specific aims in a randomized, two arm, parallel intervention of pomegranate juice or placebo for 12 weeks in obese men.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years old males (inclusive)
* BMI range from 30 to 45 (inclusive)
* Non-smokers
* Fitzpatrick Skin type II-IV
* Willing to maintain normal activity and eating patterns for the duration of the study
* Willing to maintain their normal diet for the duration of the study but avoid pomegranate products and ellagitannin rich foods.

Exclusion Criteria:

* Any subject with a history of diabetes mellitus on medications, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP>160mmHg, diastolic BP>95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
* Known cardiovascular disease, as defined by a self-reported history or medical record documentation of any of the following: myocardial infarction, angina pectoris, prior revascularization (coronary artery bypass graft, percutaneous coronary intervention), peripheral vascular disease, arrhythmias, congestive heart failure, congenital heart disease, cerebrovascular disease (stroke, transient ischemic attack).
* History of known vascular disorder or autoimmune processes including Crohn's disease, ulcerative colitis, severe psoriasis, rheumatoid arthritis, and cryoglobulinemia that may affect vascular studies.
* History of skin cancer (melanoma or non-melanoma), xeroderma, pigmetosum, systemic lupus erythematosus, or dermatomyositis.
* Any subject who is taking photosensitizing medications, i.e. Ibuprofen, Naprosyn, furosemide, hydrochlorothiazide, isotretinoin statins, and phenothizaones.
* Any subject who is taking vasoactive medications (such as nitrates, calcium channel blockers, and beta-blockers)
* Any subject with a screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
* Abnormal liver function (AST and ALT > 2 x upper limit)
* Currently taking steroidal drugs
* Cancer treated within the past two years
* Participation in a therapeutic research study within 30 days of baseline
* Use of antibiotics within one month
* Allergy or sensitivity to pomegranate products
* Follows a vegetarian, vegan or beef-free diet

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Change in erythema dose | Baseline and 12 weeks
  Assess the effect of pom juice consumption on skin resistance to UV radiation (minimal erythema dose)

SECONDARY OUTCOMES:
Change in systemic inflammation | Baseline and 12 weeks
  2. Assess the effect of pom juice consumption on systemic inflammation (serum cytokine concentration)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutriiton, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No